CLINICAL TRIAL: NCT05735301
Title: Patient Selection Based on Penumbra-core Mismatch Using MR With Non-Perfusion Imaging for Endovascular Treatment Within 6 to 24 Hours: Rationale and Trial Design
Brief Title: Patient Selection Using MR With Non-Perfusion Imaging for Endovascular Treatment Within 6 to 24 Hours
Acronym: MIELS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Director, Head of Neurosurgery, Principal Investigator, Clinical Professor, Tianjin Huanhu Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: wm-v1003
Record Dates: First submitted 2022-10-09; First posted 2023-02-21 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Endovascular Thrombectomy
Keywords: select patients; endovascular thrombectomy; magnetic resonance imaging; CT/MR perfusion; FVH-DWI mismatch
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: In this study, Patients will be screened, and image modality seletion be randomizied by a dedicated Clinical coordinator who is a non-treatment and non-follow-up participant. The randomization procedure will be computer- and web-based. Randomization is allowed when the occlusion has been established by MRA or CTA. All eligible subjects will be assigned to one of the following two treatment arms in the ratio of 1:1 after randomization:
  1. None-Perfusion group.
  2. Perfusion group.
Masking Description: The investigators will know nothing about the patient's image result until randomization. Outcome analysis was performed by an independent statistician, and results were reported directly to the data and safety regulatory committee, the investigator being aware of the results at this time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Perfusion group (Other): Non-Perfusion group consisted of patients who underwent DWI, FLAIRE, T1, and T2 sequences.The patients in the group whose MR imaging show FVH-DWI mismatch will be perfomed EVT(stent retrievers, contact aspiration, balloon angioplasty, stenting or a combination of these approaches) and best medical treatment; Patients who do not reach FVH-DWI mismatch due to image quality, EVT will be re-judged according to the DAWN criteria, Others will be given best medical treatment）
  Interventions: Procedure: Endovascular; Drug: Drug
- Perfusion group (Other): The perfusion sequence was examined by the group.The patients in the group whose F-Stroke(Brain Seal Smart Technology) indicate CBV<70mL,mismatch ratio≥1.8 mismatch Volume>15ml will be perfomed EVT and then received best medical treatment, others will be given best medical treatment only.
  Interventions: Procedure: Endovascular; Drug: Drug

INTERVENTIONS:
Procedure: Endovascular — Endovascular therapy, as an adjunct to standard stroke therapy, may be beneficial for a very select population of patients who present with an acute ischemic stroke and have a proven large, proximal occlusion on imaging.
  Endovascular therapy includes any one or more of the following:
  Intra-arterial thrombolytic therapy, aspiration, stent retrieval, or a combination of multiple mechanical devices.Remedial measures after failed thrombectomy are permitted by pharmacologic arterial thrombolysis or intravenous infusion of antiplatelet drugs, such as tirofiban or rt-PA
Drug: Drug — best drug conservative therapy could be uesd in patients who with no indication of surgery
  Other Names: Drug conservative therapy

SUMMARY:
We will conduct a multicenter, prospective, randomized, open-label, blinded endpoint trial with a non-inferiority design in patients who present 6 to 24 hours after symptom onset with LVO. Patients who meet eligibility criteria will be randomly assigned to the Non-perfusion or Perfusion group with a 1:1 ratio. In the Non-perfusion group, patients with penumbra-core mismatch (defined as the FLAIR Vascular Hyperintensity (FVH) extending beyond the boundary of the DWI cortical lesions) will receive EVT. In the Perfusion group, patients with perfusion mismatch (defined as regional cerebral blood flow (<30%) < 70 ml with mismatch ratio ≥ 1.8 and mismatch volume ≥ 15 ml) will receive EVT. Patients in both groups will receive guideline-based medical treatment. If patients in both groups do not meet the criteria for EVT, only guideline-based medical treatment will be administered.

DETAILED DESCRIPTION:
The theory of mismatch between ischemic core and penumbra has long been regarded as the triage criterion for stroke patients undergoing urgent endovascular treatment (EVT). In 1977, Astrup and colleagues first proposed the concept of ischemic penumbra through animal experiments. In 1981, Astrup defined ischemic penumbra as brain tissue surrounding the infarct core, with blood flow levels lower than those required to maintain normal brain function but higher than those causing structural changes in brain morphology . During cerebral ischemia, brain tissue exhibits a concentric distribution of varying degrees of ischemia. Tissue in the ischemic core has blood flow below 10 ml/100 g per minute and is considered irreversibly damaged. In contrast, tissue in the penumbra has blood flow between 10 and 17 ml/100 g per minute, indicating a risk of progressing to the infarct core . Patients with a high volume of penumbral tissue and a small infarct core, termed "mismatch," are deemed to derive the greatest benefit from EVT and are least likely to incur reperfusion injury risk. This principle has been consistently applied in clinical practice for stroke reperfusion, particularly in patients with late time windows, where reperfusion therapy is traditionally associated with potentially higher risks . Based on this principle, researchers utilize complex quantitative perfusion or infarct core calculation programs, often supported by artificial intelligence technology, to obtain high-quality clinical evidence. This strategy has proven successful. The efficacy and safety of EVT in patients with acute ischemic stroke (AIS) due to anterior circulation LVO is well established in multiple RCTs in the late treatment time windows (6 to 24 hours). EVT has significantly improved the prognosis of patients with LVO stroke compared to medical therapy .

DEFUSE 3 (Endovascular Therapy Following Imaging Evaluation for Ischemic Stroke 3) and DAWN (DWI or CTP Assessment With Clinical Mismatch in the Triage of Wake-Up and Late Presenting Strokes Undergoing Neurointervention With Trevo) enrolled patients showing evidence of salvageable brain tissue, determined by the presence of significant mismatch. This mismatch describes a state where the volume of viable brain tissue at risk of infarction due to ongoing vessel occlusion greatly exceeds the volume of already infarcted tissue. Mismatch evaluation used computer-generated volumetric imaging criteria, either independently (DEFUSE 3) or with clinical-core infarction criteria (DAWN) . The AURORA trial conducted a meta-analysis of data from six late-onset trials, including DAWN, DEFUSE 3, ESCAPE, REVASCAT, POSITIVE, and RESILIENT, assessing common odds ratios, favorable prognosis rates, mortality rates, and other indicators. These findings strengthen the evidence supporting the benefits of EVT for patients showing evidence of reversible cerebral ischemia within the 6-24 hour time window and are relevant to clinical practice . Detection of core infarction and penumbral mismatch is considered an effective patient screening method, capable of identifying those most likely to benefit and excluding those most likely to suffer from reperfusion injury. However, the use of urgent CTP or PWI in the emergency department is often limited in many centers worldwide . The reasons include insufficient access to appropriate technological resources, manpower requirements, and software for analyzing perfusion imaging may not be readily available. Additionally, the strict inclusion criteria based on perfusion parameters in clinical trials hinder patient selection for real-world clinical practice, leading to some patients missing the opportunity for EVT. Therefore, additional clinical and imaging criteria facilitating the identification of eligible patients would be beneficial .

In a prospective study, the presence of FVH (defined as focal, tubular, or serpentine hyperintensity in the lateral fissure, sulcus, or near the surface of the brain on the 2D FLAIR sequence) was associated with acute stroke . The exact pathophysiological mechanism of FVH remains unclear; however, its emergence suggests slow blood flow, impaired antegrade blood flow, and retrograde blood flow near the ischemic lesion . Recent research suggests that the FVH sign could serve as a significant and convenient imaging marker indicative of inadequate perfusion in patients with cerebral infarction associated with LVO. Additionally, FVH has been suggested to indirectly indicate the presence of LVO or vascular stenosis, with insufficient collateral circulation and a perfusion abnormality. The discrepancy between DWI volume and the FVH sign (FVH-DWI mismatch) in acute stroke patients could serve as a valuable penumbra-core based triage tool without the need for perfusion imaging to predict functional outcomes after stroke.

In this study, we used a randomized controlled approach to assess the risk and prognosis of EVT by identifying the presence of an ischemic penumbra using the FVH-DWI mismatch. Our aim was to establish a simple evaluation method based on the indirect assessment of penumbra-core triage without perfusion imaging on MRI to screen patients who underwent thrombolysis within 6 to 24 hours from symptom onset. We hypothesized that triage using MRI with non-perfusion imaging would be non-inferior to using perfusion imaging in demonstrating 90-day functional independence.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older；
* Anterior circulation LVO (internal carotid artery, or middle cerebral arteries (MCA)M1, M2 proximal segment) confirmed by computed tomographic angiography (CTA)/magnetic resonance angiography (MRA)；
* NIHSS score ≥6 at the time of randomization；
* ASPECTS score ≥ 6 on NCCT；
* Time from stroke onset to randomization within 6-24 hours；
* Pre-stroke mRS score 0-2；
* Completed MRI and perfusion imaging or enable to complete MRI and/or perfusion imaging；
* Signed informed consent

Exclusion Criteria:

* Pregnancy, or those potential with positive urine or serum beta Human Chorionic Gonadotrop in test；
* A history of severe allergy to contrast media；
* Uncontrolled hypertension (SBP >185mmHg; DBP>110mmHg)；
* Hereditary or acquired bleeding tendency, coagulation factor deficiency, recent anticoagulant medication (A platelet count of less than 100 x 109 /L；INR>3 or PPT more than 3 times normal)；
* Active hemorrhage or preexisting tendency to hemorrhage；
* Presence of signs of cardiac, hepatic or renal failure；
* Baseline blood glucose<50mg/dL (2.78mmol) or >400mg/dL (22.20mmol)；
* Participation in other interventional randomized clinical trials that may confound the outcome assessment of the trial；
* Life expectancy < 1 year；
* Patients who are unable to complete the 90-day follow-up；
* A stroke attack with epilepsy that prevents an accurate NIHSS score from being obtained；
* Other circumstances that the investigator considers inappropriate for participation in the trial(such as violation of guidelines or institutional processing principles during the screening process).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Functionally independent outcome in all enrolled patients | 90 days
  defined as patients with a mRS Score of 0-2 at 90 days (mRS 90d(Scores on the modified Rankin scale range from 0 to 6, with 0 indicating no symptoms, 1 no clinically significant disability, 2 slight disability, 3 moderate disability, 4 moderately severe disability, 5 severe disability, and 6 death,) of a randomized group of modified intention-to-treat (mITT) patients (defined as patients with acute macrovascular occlusions treated optimally with endovascular or pharmacologic therapy) at 90 days (with an assessment time window of ±14 days) and analyzed for noninferiority.

SECONDARY OUTCOMES:
Modified Rankin scale scores at 90 days | 90 days
  (mRS 90d(Scores on the modified Rankin scale range from 0 to 6, with 0 indicating no symptoms, 1 no clinically significant disability, 2 slight disability, 3 moderate disability, 4 moderately severe disability, 5 severe disability, and 6 death,) of a randomized group of modified intention-to-treat (mITT) patients (defined as patients with acute macrovascular occlusions treated optimally with endovascular or pharmacologic therapy) at 90 days (with an assessment time window of ±14 days) and analyzed for noninferiority.
Successful reperfusion after endovascular treatment | immediately the surgeon thought the thrombectomy completed and performed a second cerebral angiography
  extended Thrombolysis in Cerebral Infarction (eTICI) score of 2b, 2c or 3.
Recanalization rate | 72 hours
  Number of subjects who achieved successful reperfusion/total number of subjects who received endovascular treatment, confirmed by MRA, CTA, or digital subtraction angiography (DSA).
Final infarct volume | 72hours
  change from baseline in the infarct volume as calculated by CBF or DWI.
NIHSS score | 24 hours、72hour sand 7 days postoperatively
  scores range from 0 to 42, with higher scores indicating a more severe deficit.
Quality of life assessment at 90 days | 90 days
  European Five Dimensions and Five Levels Scale (EQ-5D-5L) scores (range, -0.39 [worst] to 1.00 [best]); Barthel Index scores at 90 days (range, 0 [severe disability] to 100 [no disability]).
mortality | 90 days
  mortality of all-cause.
symptomatic intracranial hemorrhage | 48 hours
  the presence of extravascular blood in the cranium that was associated with an increase in the NIHSS score of ≥4 points or death and was judged to be the predominant cause of neurologic deterioration.
FVH-ASPECT score | 24 hours、72hour sand 7 days postoperatively
  FVH-ASPECTS: 0-7, with 0 indicating absence of FVH and 7 suggesting prominent FVH

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wei, doctorate, Principal Investigator — Tianjin Huanhu Hospital
Locations (1):
- TianJinHH, Tianjin, Tianjin Municipality, China